CLINICAL TRIAL: NCT01714934
Title: Study of Pepsin Levels in the Broncho-Alveolar-Lavage Fluid of Patients With Idiopathic Pulmonary Fibrosis
Brief Title: The Role of Gastric Content Microaspirations in the Pathogenesis of Idiopathic Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9440-TS-CTIL
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: IDIOPATHIC PULMONARY FIBROSIS
Keywords: IDIOPATHIC PULMONARY FIBROSIS; MICROASPIRATION
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: BAL broncho alveolar lavage at bronchoscopy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IPF: IPF patients diagnosed according to clinical and radiological findings
- NON IPF: Other interstitial lung diseases such as sarcoidosis or hypersensitivity pneumonitis diagnosed as per clinical and radiological findings

SUMMARY:
The pathogenesis of idiopathic pulmonary fibrosis (IPF) is debatable. Looking for an insult to lung parenchyma that generates the pathogenesis of the disease is challenging. Pepsin is a proteolytic enzyme present in the gastric juice. Microaspirations of gastric content were described as a potential factor for injury in many chronic lung disorders. Bronchoalveolar lavage (BAL) is a routine investigation technique in interstitial lung diseases. The presence of pepsin in the BAL fluid recovered from patients with IPF may indicate a possible role for gastric microaspirations in the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with interstitial lung disorders including IPF

Exclusion Criteria:

* patients younger than 18 years or older than 85,
* pregnant women,
* patients that present with medical conditions contra -indicated for performing bronchoscopy including sedation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPF versus patients with other interstitial lung disorders (non IPF)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
BAL Pepsin level | 18 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel